CLINICAL TRIAL: NCT06107140
Title: Duration of Dual Antiretroviral Therapy in Virologically Suppressed People Living With HIV and Factors Associated With Switching to Tritherapy : a Real-life Cohort
Acronym: TOBIT
Status: Completed | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHT/URC/2023/13
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: HIV Infections
Keywords: epidemiology
MeSH Terms: conditions — HIV Infections | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dual therapy — The evaluation will focus on the retention of patients living with hiv on dual antiretroviral therapy.

SUMMARY:
HIV infection requires lifelong continuous antiretroviral (ARV) treatment. The efficacy of current ARV treatments makes it possible to propose strategies for reducing the cumulative exposure to ARVs, side effects and costs. And so improve the quality of life of people living with HIV (PLHIV). However, in the real world, less regular adherence to treatment, more heavily pre-treated patients and resistance to treatment make these dual therapies prescribed beyond the strict framework of clinical trials. This can lead to undesirable side effects. From the perspective of personalized medicine, it seems to be important to determine which patients are receiving dual ARV therapy, and which patients remain on it for a long time. Identifying prognostic factors would enable us to adapt therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* hiv patient
* viral load < 50copies/ml
* patient treated with dual therapy
* patients with hospital follow-up between 2011 and 2023

Exclusion Criteria:

* adults under legal protection
* underage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed up in a referral center for the management of PLHIV who started dual antiretroviral therapy in the period from 2011 to 2023 and whose viral load was < 50 copies/ml before initiation of dual therapy.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
therapeutic switch | 5 years
  Proportion of patients switching from dual to triple therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier DRON, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No